CLINICAL TRIAL: NCT04998734
Title: ASI-SR Form as a Standardized Instrument for Healthcare Management of Chronic Non-cancer Pain Patients
Brief Title: Validation of the ASI-SR Form in a Population of Chronic Non-cancer Pain Patients
Acronym: ASI-SR
Status: Terminated | Type: Observational
Why Stopped: Recruitment failure
Sponsor: Uppsala University (Other)
Collaborators: Uppsala University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2020-001-5
Record Dates: First submitted 2021-08-02; First posted 2021-08-10 (Actual); Last update posted 2023-05-11 (Actual); Status verified 2023-05

CONDITIONS: Chronic Pain; Opioid-use Disorder; Quality of Life; Risk Reduction; Assessment, Self
Keywords: opioids; ASI-SR; pain; opioid-use disorder; dependence; validation; assessment
MeSH Terms: conditions — Chronic Pain; Opioid-Related Disorders; Risk Reduction Behavior; Pain

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Chronic pain: Patients with chronic non-cancer pain referred to secondary and tertiary care
  Interventions: Diagnostic Test: ASI-SR

INTERVENTIONS:
Diagnostic Test: ASI-SR — Psychometric properties of ASI-SR

SUMMARY:
The Swedish version of ASI-SR has shown good feasibility in assessment of addiction patients functioning compare to long and time-consuming ASI, which is upp to date golden standard in Sweden. This study investigate if ASI-SR is suitable instrument for the assessment of the chronic pain patient addicted to opioids. The validation process is designed according to the COSMIN guidelines.

Preliminary results are expected by December 2022.

DETAILED DESCRIPTION:
The use of opioids in treatment of chronic non- cancer pain (CNCP) has increased during the past decades in most parts of the western world. Use of prescription opioids can lead to problematic opioid use which can be life-threatening with significant morbidity and mortality. Studies have found that 21-29% of CNCP patients receiving chronic opioid therapy (COT) ( receiving opioids for > 90 days) have problematic opioid use. Individuals with chronic pain and co-occurring substance use disorders and/or mental health disorders, have increased risk for problematic use of prescribed opioids.

Several screening instruments and strategies have been introduced in recent years for identifying patients not suitable for opioid therapy. Even so, there is no single test or instrument that can reliably identify those patients at risk for developing problematic opioid use or opioid use disorder if opioid therapy is initiated, or identify those who need increased monitoring during treatment.

Addiction Severity Index (ASI) is a standardized semi-structured interview used for assessing severity and need of treatment in seven functional domains associated to substance use disorders; physical health, employment/support status, alcohol use, drug use, legal status, family/social functioning and psychiatric health. The ASI was developed in the US. by McLellan and colleagues and is widely used all over the world, both in research and for clinical assessment and treatment evaluations . The ASI could be a useful instrument for a multidimensional assessment of patients with chronic non-cancer where opioid treatment is considered, and it could also be used for evaluation of ongoing opioid therapy . However, the ASI interview is a time consuming instrument. To conduct an interview takes between 45-60 minutes and is followed by 20-25 minutes of administrative work. In the year of 2000 Rosen et al tested a short self-report form based the items used to calculate the ASI composite scores that asses current function and problem severity. This questionnaire was translated by our research group and tested on a sample of individuals referred to the Addiction clinic at Uppsala University Hospital. The study suggested that a self-administered questionnaire based on the subscales of the ASI composite scores is a feasible alternative to the ASI interview for assessing patient functioning in the different domains and screen for current problematic alcohol- or drug use .

A validated screening tool that provides both an effective method of assessing patients and identifying problems in several different life domains, and identify substance use related problems if they should arise, would be beneficial in clinical practice when deciding what treatment to offer. Such an instrument could potentially decrease the risk of iatrogenic opioid use disorder.

Purpose and aims The main objective with this study is to test the psychometric properties of the ASI-SR in a population of CNCP patients. 'Secondary aim is to describe differences between subjects treated within the substitution therapy program and those who are treated within the pain clinic.

Method:

Sample Participants for this study will be recruited from outpatient pain clinic and addiction clinic at Uppsala University Hospital, and Linköping University Hospital Sweden. Eligible for participation are persons >18-65 years of age with current CNCP and ongoing treatment at the facilities. Estimated number of participant needed is about 200.

Exclusion criteria are severe cognitive impairment, illiterate in Swedish, and inability to give informed consent.

Procedures Eligible participants will be approached and asked if they can consider to participate in the study by clinical staff at the facilities. If they accept, they will receive an e-mail with a link to the questionnaires and to written information about the study. If they decide to participate they will give informed consent by signing a digital consent form. A digital battery of questionnaires containing the ASI-SR and a validity battery will then be provided to the participants to fill out. The validity battery will consist of self-report forms. To participants that do not respond to the questionnaires and have not declined participation, reminders will be sent out by text-messages, e-mail and mail. Four days after the participants have completed the questionnaires they will receive an e-mail with a link the ASI-SR form to fill out once more to test re-test reliability.

Participants that do not want to or do not have access to the digitalized versions of the questionnaires will be offered to fill out paper versions of the questionnaires sent to them by mail.

Measures ASI-SR is a 38 question self-administered form based on the items used to calculate the ASI's composite scores, measuring current problems and severity in seven domains . The CS ranges from 0 to 1 where 0 indicates no problems.

The validity battery consist of self-administered questionnaires that correspond to six out of seven of the ASI-SR's domains. These questionnaires will be used as concurrent validity measures for all the ASI-SR composite scores (CS) except the CS for legal situation. The participants will fill out questions about current pain intensity and pain interference, the Rand 36 for multidimensional health related quality of life , pain related disability Pain Disability Index (PDI) and Sheehan Disability Scale (SDS) which measures disability across domains of work/school, social life, and family life/home responsibilities . The Alcohol Use Disorder Identification Test (AUDIT) will be used for assessment of problematic alcohol use and the Drug Use Disorder Identification Test (DUDIT) for assessment of problematic illicit drug use . PHQ9 will assess depressive symptoms and the GAD 7 will be used for assessment of anxiety symptoms . Patient global impression of change (P-GIC) will be used to evaluate if the participants experienced any changes in global health between test-retest of the ASI-SR. P-GIC is gold standard for measuring change in CNCP patients .

Statistics Statistical analyses will be done using SPSS (Version 23, IBM SPSS Statistics for Windows, Armonk, NY: IBM Corp). Calculation of the CS follow standard procedure . Consistency of CS between the interview and the self-report will be evaluated on the individual basis by interclass correlation analysis (ICC) and at group level with paired t-test or Wilcoxon signed rank test if data is not normally distributed. ICC coefficient is considered to be poor if it is less than 0.40, fair between 0.40-0.59 , good between 0.60-0.70 and excellent between 0.75-1.00 .

Reliability and internal consistency will be evaluated using Cronbach's α. The α coefficient is considered acceptable if it is above 0.70 .

The concurrent validity of each score will be assessed with suitable correlation analyses between the ASI-SR composite score(s) and the external validity measure(s).

To assess discriminant validity of the ASI-SR composite scores and external validity measures, an intercorrelation matrix between ASI-SR composite scores, and composite scores and external measures will be computed.

For evaluating factor structure principal component analyses (PCA) will be used.

Relevance for the field Opioid therapy for chronic non-cancer pain has emerged as a problematic treatment and the evidence is scarce for its effectiveness . However, there are some individuals that seem to benefit from opioid therapy and most guidelines propose an individual approach to management, beginning with a comprehensive patient evaluation, focusing on factors that may indicate potential substance use disorder. When opioids are used, clinicians should closely monitor patients for loss of response, adverse effects or aberrant behavior, and assess treatment outcome . There is a need for a multi-dimensional instrument that can assess problems related to increased risk for developing problematic opioid use, i.e. opioid use disorder, psychiatric co-morbidity and social problems. The ASI-SR could be an effective way of screening for current problems in different life domains and to monitor and evaluate ongoing treatment and identify problems if they would arise. Additional measures include urine or saliva drug testing, prescription practice, opioid treatment agreements, and universal precautions in conjunction with opioid therapy.

Ethical considerations The study will be sent to the Regional Ethical Review Board in Uppsala. Participants will be anonymous and all data will be coded before processed.

ELIGIBILITY:
Inclusion Criteria:

* Chronic non-cancer related pain
* ongoing treatment in the clinic

Exclusion Criteria:

* severe cognitive impairment
* illiterate in Swedish
* inability to give informed consent.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: In this days there are approx. 100 patients treated in the substitution program, 1300 patients receiving referral to the pain clinic in Uppsala Pain Center.
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2021-08-05 (Actual); Primary Completion 2022-06-01 (Actual); Study Completion 2023-03-28 (Actual)

PRIMARY OUTCOMES:
Addiction Severity Index - Short version | Baseline
  The main objective with this study is to test the psychometric properties of the ASI-SR in a population of CNCP patients.Consistency of CS between the interview and the self-report will be evaluated on the individual basis by interclass correlation analysis (ICC) and at group level with paired t-test or Wilcoxon signed rank test if data is not normally distributed. ICC coefficient is considered to be poor if it is less than 0.40, fair between 0.40-0.59 , good between 0.60-0.70 and excellent between 0.75-1.00.

SECONDARY OUTCOMES:
Patient Global Impression of Change | Baseline
  7-grade scale (-3-+3)where the lowest points indicate negative and highest points indicate positive change.
Addiction Severity Index -Short version | 4-7 days later
  Second test ASI-SR for reproducibility( 0,1 answer /scores in different categories)
Generalised Anxiety Disorder 7 | baseline
  Generalised Anxiety Disorder 7-item scale (0-21) The higher the score the higher severity of the anxiety disorder, cut-off 10.
Research and Development 36-Item Health Survey RAND-36 | Baseline
  Quality of life instrument of International Resource Center for Health Care considering both physical and mental health aspects. Scores 0-100. The Higher score the better quality of life in different segments of well-being, function or quality of life.
Pain Disability Index | Baseline
  7-question score system for different pain groups,(0-70). The higher the index the greater the persons disability due to the pain.
Alcohol Use Disorder Identification Test | Baseline
  Scoring system, (0-40)where increase of the points reflects increased risk of problematic alcohol use.
Drug Use Disorder Identification Test | Baseline
  Scoring system,(0-44) where increase of the points reflects increased probability of drug abuse syndrome.
Patient Health Questionnaire PHQ9 | Baseline
  Depression Assesment scoring system, (0-15) where <4 is no need of depression treatment, and >15 identifies need of pharmacologic or other depression treatment

OTHER OUTCOMES:
Descriptive characteristics of the group | Baseline
  Age, sex, educational level, occupational status etc For evaluating factor structure principal component analyses (PCA) will be used.

CONTACTS AND LOCATIONS:
Overall Officials: Pernilla Åsenlöf, Profesor, Principal Investigator — Uppsala University
Locations (1):
- Uppsala University Hospital, Pain Center, Uppsala, Sweden

IPD SHARING:
Plan to Share IPD: No